CLINICAL TRIAL: NCT02112266
Title: Online Assessment for Therapy Expectation and Quality of Life and Online Therapy of Depression
Brief Title: Depression Online Assessment and Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Makora (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ICBT; 2013-0542 (Other: KEK Zurich CH)
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: depression; online therapy; cognitive behavioural therapy; quality of life; alexithymia; therapy expectation and satisfaction
MeSH Terms: conditions — Depression; Affective Symptoms; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no mail support (Other): no mail support during follow-up
  Interventions: Other: no mail support
- mail support (Other)
  Interventions: Other: Mail support

INTERVENTIONS:
Other: Mail support — between post treatment and follow up two groups: one with unspecific mail support every 2 weeks one without
  Arms: mail support
Other: no mail support — follow-up without mail support
  Arms: no mail support

SUMMARY:
One Aim of the current study is to better understand why some patients suffering from depression do not seek professional help by doctors but in the internet.

Furthermore patients with depression will receive Online Therapy for depression. Aim of this part of the study is to investigate whether quality of life changes accordingly to improvement of symptoms after online therapy.

DETAILED DESCRIPTION:
* German speaking patients can register online. There will be no side visits.
* After screening: patients which meet inclusion criteria and no exclusion criteria can take part in online therapy for depression.
* After 12 weeks 2nd online survey. After this survey patients can use the program the following 6 months (follow-up)
* After 6 months 3rd and last online-survey.
* According to the aims of the study cross-sectional as well as longitudinal data will be obtained and analysed

ELIGIBILITY:
Inclusion Criteria:

* German language
* depression at least slight according BDI (Beck depression inventory) and at least 2 weeks

Exclusion Criteria:

* severe depression according BDI
* suicidal ideation
* alcohol or drug dependency
* history of psychotic symptoms
* history of bipolar disorder or previous mania
* current in-patient care or semi-residential treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change of Quality of life | at screening, post treatment (3 months) and follow-up (6 months after post)
  WHOQol brev - WHO quality of life questionnaire short form

SECONDARY OUTCOMES:
change of Sleep quality | screening, post treatment (3 months), follow-up(6 months after post)
  Questionnaire PSQI - Pittsburgh sleep quality index
change of severity of depression | 3 time points screening, + 3 months + 6 months
  patients receive mail support or not during follow up. Questionnaire: BDI - Beck Depression Inventory

OTHER OUTCOMES:
change of therapy expectation during online-therapy | 3 time points screening + 3 months + 6 months
  therapy expectation at screening and after intervention. Questionnaire: PECHI - Psychotherapy Expectations, Concerns, and Hopes Inventory
alexithymia | screening
  influences on outcome? Questionnaire: TAS - Toronto Alexithymia Scale
satisfaction with current and former therapies and influence on decision for online therapy | screening
  adapted version of ZUF-8 (= "Zufriedenheitsfragebogen mit der Behandlung" english version CSQ- client satisfaction questionnaire) for different experiences with therapy (e.g. for depression, for other psychiatric illnesses)
sense of coherence | screening
  influencing outcome? measured with SOC-13 -Sense of Coherence Scale
changes in sense of coherence | + 3 months after screening (post) and + 6 months after post
  measured with SOC-13 does online-therapy helps to develop a better SOC?
changes alexithymia | + 3 months after screening (post) , + 6 months after post
  Trait and state characteristics of alexithymia in depression measured with TAS-20

CONTACTS AND LOCATIONS:
Overall Officials: S Weidt, MD, Principal Investigator — USZ, UZH
Locations (1):
- University Hospital Zurich - only online recruitment, Zurich, Canton of Zurich, Switzerland